CLINICAL TRIAL: NCT03540511
Title: Prognostic Value of Postoperative Troponin in Patients With Renal Dysfunction Undergoing Cardiac Surgery
Brief Title: Postoperative Troponin in Renal Dysfunction After Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Youn Joung Cho, MD, Clinical assistant professor, Seoul National University Hospital
Other Study IDs: TnI_CKD
Record Dates: First submitted 2018-05-15; First posted 2018-05-30 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Renal Dysfunction
Keywords: cardiac surgery; troponin; mortality
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: postoperative troponin — assess postoperative troponin levels after cardiac surgery in patients with renal dysfunction

SUMMARY:
Elevated level of troponin is frequently observed among patients with renal dysfunction. Increase in troponin after cardiac surgery may predict postoperative outcome in cardiac surgery patients. However, the relationship between the increased troponin and outcome after cardiac surgery has not been fully elucidated in patients with renal dysfunction.

DETAILED DESCRIPTION:
This is a retrospective observational study to evaluate the prognostic value of postoperative troponin in patients with renal dysfunction undergoing cardiac surgery. Electrical medical records of patients who underwent cardiac surgery between 2004 and 2015 will be assessed. Perioperative laboratory data including troponin and glomerular filtration rate, type of surgery, and outcome variables including mortality will be analysed to determine the prognostic value of postoperative value of postoperative troponin in patients with renal dysfunction undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with renal dysfunction who underwent cardiac surgery between 2004 and 2015 at Seoul National University Hospital

Exclusion Criteria:

* Patients without laboratory information on glomerular filtration rate or troponin levels

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with renal dysfunction who underwent cardiac surgery between 2004 and 2015 at Seoul National University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
mortality | through study completion, average 3 years
  mortality after cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Youn Joung Cho, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided